CLINICAL TRIAL: NCT06528938
Title: Randomized Pilot Trial Comparing the Feasibility and Efficacy of Accelerated vs. Standard fMRI-guided iTBS in Treatment-Resistant Depression in Adolescents
Brief Title: Comparing the Efficacy of Accelerated vs. Standard fMRI-guided iTBS in Treating Adolescents Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Sara Tremblay, Principal Investigator, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0047
Record Dates: First submitted 2024-06-14; First posted 2024-07-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Depression; Depressive Disorder, Major
Keywords: Accelerated rTMS; repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accelerated iTBS (Active Comparator): Intermittent Theta Burst Stimulation (iTBS) will be applied to the left dorsolateral prefrontal cortex (DLPFC). Participants will receive daily sessions (Mon-Fri), three times a day for 10 days (2 weeks).
  Interventions: Device: Theta Burst Stimulation
- Standard iTBS (Active Comparator): Intermittent Theta Burst Stimulation (iTBS) will be applied to the left DLPFC. Participants will receive daily sessions (Mon-Fri), once a day for 30 days (6 weeks).
  Interventions: Device: Theta Burst Stimulation

INTERVENTIONS:
Device: Theta Burst Stimulation — Cool B70 coil (left DLPFC) with X100 MagPro rTMS Device (Magventure A/S, Farum, Denmark)

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a Health Canada approved treatment for major depression. Theta burst stimulation (TBS), a type of rTMS, is a very promising new treatment for major depression in adults and adolescents. However, very few studies have assessed the efficacy of accelerated, three times a day TBS in comparison with standard once a day TBS in adolescents. The study aims to explore further evidence in hopes to conduct a large-scale, randomized, multisite, placebo-controlled clinical trial evaluating the effects of a functional magnetic resonance imaging (fMRI)-guided accelerated rTMS protocol vs. standard once/daily rTMS for treatment-resistant depression in adolescents.

DETAILED DESCRIPTION:
Recently the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) has significantly improved for Treatment-Resistant Depression (TRD) in adults and promising evidence suggesting safety and efficacy of rTMS in adolescents. These youth studies currently use outdated stimulation protocols, with most of them using treatments on a once/daily schedule. Given the prevalence, morbidity, and mortality associated with depression in adolescents, and considering that over 40% of adolescents do not respond to medications, a randomized controlled trial (RCT) to establish the safety and efficacy of new rTMS protocols for difficult-to-treat depression in adolescents is desperately needed.

This open-label randomized controlled trial will compare accelerated intermittent theta burst stimulation (iTBS) and standard once a day iTBS in adolescents with major depressive disorder (MDD). For this pilot trial, 10 adolescents (5 females, 5 males) with treatment-resistant depression will be recruited. Each participant will undergo a 30-40-minute magnetic resonance imaging (MRI) scan, after which they will receive iTBS applied to the left dorsolateral prefrontal cortex (DLPFC) once a day for 6 weeks (standard treatment) or for an accelerated duration of 3 times a day for 2 weeks. Symptoms will be assessed through clinical assessments as well as self-report questionnaires. Prior to treatment start each participant will complete the clinical assessments as well as the self-report questionnaires for a baseline measurement. The self-report measures will be completed every 5th treatment (total of 7 times including baseline). The clinical assessments will be completed after the 15th and 30th treatment, as well as 2-,4-, and 12-weeks post treatment course (total of 6 times including baseline). The main outcome of this trial is a clinical response rate which will be defined as a ≥ 50% reduction in depressive symptoms based off of the Children's Depression Rating Scale Revised for depression (CDRS-R). The secondary outcome of this trial is suicidal ideation which will be measured by the Beck Scale for Suicidal Ideation (BSS), as well as several other outcomes such as anxiety, sleep quality, physical activity and stress. The ultimate goal of this study is to provide initial evidence for conducting a large-scale, randomized, multisite, placebo-controlled clinical trial evaluating the effects of an fMRI-guided accelerated rTMS protocol vs. standard once/daily rTMS for treatment-resistant depression in adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and competent to consent.
2. Ages 16-19 years old.
3. Can speak and read English.
4. Primary and/or predominant diagnosis of major depressive episode without psychotic features in the current episode, confirmed by The Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
5. Depressive symptoms have not improved after ≥ 1 adequate dose of antidepressant in the current depressive episode.
6. Moderate symptoms in the current depressive episode, indexed by a score of at least 40 on the Children's Depression Rating Scale Revised for depression (CDRS-R).
7. Are able to adhere to the treatment schedule.
8. Have stable psychotropic medications and/or psychotherapy regimen for at least four weeks before participating in the trial.

Exclusion Criteria:

1. Diagnosis of bipolar I or II disorder, based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.
2. Current or past substance (< 3 months) (excluding caffeine or nicotine) or alcohol abuse/dependence, as defined in the DSM-5 criteria. Based on DSM-5 criteria, mild cannabis or alcohol use would be allowed in the past 3 months, moderate to severe would be an exclusion.
3. Current use of illegal substances or cannabis confirmed by urine screening test.
4. Concomitant unstable major medical or neurological disease (e.g., uncontrolled diabetes or renal dysfunction).
5. Organic cause of depressive symptoms (e.g. thyroid dysfunction), ruled out by the treating physician.
6. Acute suicidality or life-threatening due to self-neglect.
7. Are pregnant or breastfeeding, or plan to become pregnant during treatment (pregnancy will be assessed by a urine test).
8. Have a specific contraindication to TMS and/or MRI (e.g., personal history of epilepsy or seizures, metal head implant, pacemaker).
9. Unwilling to maintain the current antidepressant regimen.
10. Taking more than 1 mg/day of lorazepam or equivalent.
11. Any other condition that, in the opinion of the investigators, would impair the participant's ability to complete the study.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Compare the efficacy of accelerated intermittent theta burst stimulation (iTBS) and standard once daily iTBS on clinical response in adolescents. | Administered at screening, weekly for 2 weeks in accelerated group, every 3rd week for 6 weeks in once/daily (standard) group, as well as 2-, 4- and 12-weeks post-treatment course for both treatment protocols.
  Clinical response will be defined as a ≥ 50% reduction in depressive symptoms based on the Children's Depression Rating Scale Revised for depression (CDRS-R). The CDRS-R is a clinician-evaluated instrument consisting of 17 items used to measure the severity of depressive episodes in a pediatric population in children 6 to 12 years of age that has been shown to be applicable in adolescents as well. The overall score ranges from 17 to 113, where scores of ≥40 suggest moderate to severe depression and ≤28 is defined as remission or asymptomatic. In this study, a response to treatment will be defined as a reduction of 50% or more on the overall CDRS-R score at the post-intervention assessment (post-treatment 30).

SECONDARY OUTCOMES:
Change in self-reported suicidal ideation as measured by Beck Scale for Suicidal Ideation (BSS). | Administered at screening, every other day for 2 weeks in accelerated group, weekly for 6 weeks in once/daily (standard) group, as well as 2-, 4- and 12-weeks post-treatment course for both treatment protocols.
  The BSS is a self-administered questionnaire consisting of 19 items that assesses an individual's presence of suicidal ideations and intensity. Each item is rated on a scale of 0 to 2, with a possible total score ranging from 0 to 38. Several other questionnaires addressing anxiety, sleep quality, physical activity and stress, among others, will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tremblay, PhD, Principal Investigator — The Royal's Institute of Mental Health Research; Jean-François Lepage, PhD, Principal Investigator — Sherbrooke University
Locations (1):
- The Royal's Institute of Mental Health Research, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data collected from this study (IPD) will be de-identified for all parties who have permission to access it. This de-identified data may be shared with other researchers at the Royal's Institute of Mental Health Research. De-identified may be shared with the public only upon request. Please note that all data that has the potential of revealing participants' identity will NOT be used to shared.
Supporting Information: SAP
Time Frame: De-identified data may become available (upon request) when the study is completed and published (anticipated time frame: the year of 2026)
Access Criteria: De-identified data will be accessible only through the permission of the lead research scientist. All requests must be made and accepted by her.